CLINICAL TRIAL: NCT00958659
Title: Prognostic Multigene Expression Classification of Neuroblastoma Patients
Brief Title: Study of Specimens From Young Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL08B1; NCI-2011-02190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-NB-2008-01 (Other: Children's Oncology Group); ANBL08B1 (Other: CTEP); COG-ANBL08B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Regional Neuroblastoma; Stage 4S Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (gene expression profiling): Previously collected samples are analyzed for 59 prognostic genes by real-time quantitative PCR-based gene expression profiling.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies specimens from young patients with neuroblastoma. Studying the genes expressed in specimens from patients with cancer may help doctors identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish a robust messenger ribonucleic acid (mRNA) gene expression classifier for improved outcome prediction in children with neuroblastoma by using real-time polymerase chain reaction (PCR) to quantify mRNA levels from genes that have been shown in at least 2 independent studies to have predictive power.

II. Identify microRNA (miRNA) patterns that have prognostic significance in neuroblastoma (NB) as accumulating evidence indicates that alterations in miRNA expression play a critical role in tumorigenesis and can be used in prognostic evaluation.

III. To perform an integrated analysis of the established microRNA classifier with our mRNA signature to determine whether it results in even better classification of NB tumors.

OUTLINE:

Previously collected samples are analyzed for 59 prognostic genes by real-time quantitative PCR-based gene expression profiling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Neuroblastoma

  * Untreated disease
* RNA samples from primary untreated NB-tumors available in Children's Oncology Group (COG) repository

  * At least 60% tumor cells
* At least 2 years of follow-up from the date of diagnosis
* Full clinical and biological annotation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With Neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2008-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
mRNA expression levels from genes that have been shown (in at least two independent studies) to have power for outcome prediction in children with NB, assessed by real-time PCR | Baseline
  Multivariate logistic regression analyses will be performed to determine if the mRNA expression signature is a significant independent predictor after controlling for currently used risk factors.
miRNA patterns that have prognostic significance in NB, assessed by a reverse transcription quantitative PCR-based 'stem-loop' method to quantify expression levels | Baseline
  Multivariate logistic regression analyses will be performed to determine if the miRNA expression signature is a significant independent predictor after controlling for currently used risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hogarty, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States